CLINICAL TRIAL: NCT01167205
Title: Positive Effects of Haematococcus Astaxanthin on Oxidative Stress and Lipid Profile in Overweight and Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: C-1005-072-319
Record Dates: First submitted 2010-07-08; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Healthy; Overweight; Obesity
Keywords: Healthy adults with BMI over 25.0 kg/m2
MeSH Terms: conditions — Overweight; Obesity | interventions — astaxanthine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: astaxanthin — astaxanthin 20mg for 12 weeks

SUMMARY:
The purpose of this study is to determine whether astaxanthin (ASX) supplementation will reduce obesity-induced oxidative stress and improve lipid profile in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with BMI over 25.0 kg/m2
* Non-smoker

Exclusion Criteria:

* Excessive alcohol consumption
* Pregnant or lactating women
* Dyslipidemia, hyperglycemia, or other chronic diseases.
* Subjects who were taking vitamin supplements

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2010-08; Primary Completion 2010-12; Study Completion 2011-03

PRIMARY OUTCOMES:
Evaluation of the plasma MDA (malonaldehyde) level | 12 weeks
  MDA is a three chain aldehyde produced during the composition of a lipid hydroperoxide and is a well known indicator of lipid peroxidation.
  The purpose of this stduy is to determine whether ASX supplementation lowers oxidative stress using MDA,a biomarker.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute Seoul National University Hospital, Seoul, Seoul, South Korea